CLINICAL TRIAL: NCT04716257
Title: Impact of Different Treatment Strategies on the Prognosis of Ovarian Metastatic Colorectal Cancer Patients: a Prospective, Multi-center, Real-world Study
Brief Title: A Prospective, Multi-center, Real-world Study of Ovarian Metastatic Colorectal Cancer Patients
Acronym: proOMCRC
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: Sun Yat-sen University (Other); Cancer Hospital of China Medical University, Liaoning Cancer Hospital & Institute (Unknown); Changhai Hospital, Naval Medical University (Unknown)
Responsible Party: Principal Investigator, Meng Qiu, Prof., West China Hospital
Other Study IDs: 20201296
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Metastasis; Colorectal Cancer
MeSH Terms: conditions — Krukenberg Tumor; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — samples of ovarian metastases if available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, multi-center, real-world study is conducted to investigate the impact of different treatment strategies (systemic chemotherapy combined with oophorectomy or with other local treatment or chemotherapy alone) on the prognosis of ovarian metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
This study prospectively collects data of patients diagnosed with ovarian metastatic colorectal cancer, meeting inclusion criteria and signing the informed consent. Patients' treatment strategies and survival outcome in the real world will be faithfully recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal adenocarcinoma;
2. Histologically or radiologically diagnosed with ovarian metastasis, whether or not combined with metastases in other organs;
3. Women ≥18 years of age;
4. Eastern Cooperative Oncology Group performance status score ≤2;
5. Available imaging data if the disease is measurable according to RECIST criteria version 1.1; patients are eligible if there is no measurable lesion.
6. Complete medical records;
7. Informed consent form signed.

Exclusion Criteria:

1. Not ovarian metastatic colorectal cancer confirmed by radiology or histology;
2. Drug abuse or other medical, psychological and social disorders that would interfere with cooperation with the requirements of the study;
3. Other conditions that would influence patient compliance;
4. Pregnant or breastfeeding female; male and female unwilling to take any contraceptive measures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ovarian metastatic colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Ovarian specific overall survival | up to 3 years
  Calculated from the date of diagnosis with ovarian metastasis to death (caused by cancer) or last follow-up time.

SECONDARY OUTCOMES:
Ovarian specific objective response rate | 6 months
  Response rate of ovarian metastases to systemic chemotherapy
Extra-ovarian specific objective response rate | 6 months
  Response rate of extra-ovarian metastases to systemic chemotherapy
Progression free survival | 6 months
  Survival time from treatment start to disease progression or death.
Quality of life questionnaire | 6 months
  Quality of life during treatment

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital of China Medical University, Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Changhai Hospital, Naval Medical University, Shanghai